CLINICAL TRIAL: NCT01113099
Title: Assisted Detailing to Improve Guideline Adherence
Brief Title: Improving Adherence to Prescribing Guidelines for Cholesterol Lowering in Hospitalized Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Thomas C Bailey/Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 02-1072; R01HL070790 (NIH)
Record Dates: First submitted 2010-04-22; First posted 2010-04-29 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2010-04

CONDITIONS: Diabetes; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Academic detailing of physicians (Experimental)
  Interventions: Other: Academic detailing
- Usual care (No Intervention)

INTERVENTIONS:
Other: Academic detailing — Education of physicians by pharmacists regarding indications for statins in diabetic patients
  Arms: Academic detailing of physicians

SUMMARY:
We hypothesize that when compared to usual care a greater proportion of hospitalized diabetic patients who are candidates for cholesterol lowering will be discharged with a prescription for a statin if their physicians are contacted by a pharmacist to discuss treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with diabetes
* LDL >= 100

Exclusion Criteria:

* Terminal illness
* Pregnancy
* Intolerance or contraindication to statin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Statin prescription at hospital discharge | Hospital discharge (avg = 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Bailey, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Result] McKinnon PS, Seaton T, Noirot LA, Reichley RM, Heard KM, Shannon WD, Goldberg AC, Dunagan WC, Bailey TC. Improving adherence to dyslipidemia medication guidelines in hospitalized diabetic patients using a technology-assisted pharmacist intervention. AMIA Annu Symp Proc. 2008 Nov 6:868. PMID 18999065
- [Result] Reichley R, McKinnon PS, Seaton T, Noirot L, Dunagan WC, Bailey TC. Adherence to dyslipidemia treatment guidelines in diabetic patients. AMIA Annu Symp Proc. 2006;2006:1071. PMID 17238690
- [Result] Reichley R, Rachmiel E, Seaton T, Noirot L, Longyhore D, Dunagan WC, Bailey TC. Intervention to improve dyslipidemia screening in hospitalized diabetics. AMIA Annu Symp Proc. 2005;2005:1093. PMID 16779380
- [Result] McKinnon PS, Reichley RM, Noirot LA, Dunagan WC, Bailey TC. Prospective validation of an algorithm to identify hospitalized diabetic patients using administrative data. AMIA Annu Symp Proc. 2006;2006:1029. PMID 17238648